CLINICAL TRIAL: NCT06923267
Title: Ultrasound Evaluation of Cardiac Function During Three Spontaneous Breathing Trials in Intensive Care Unit : A Prospective Interventional Study
Brief Title: Ultrasound Evaluation of Cardiac Function During Spontaneous Breathing Trials
Acronym: ATARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUO-2024-09
Record Dates: First submitted 2025-03-10; First posted 2025-04-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Weaning Invasive Mechanical Ventilation; Weaning-induced Pulmonary Edema; Weaning Failure of Mechanical Ventilation; Spontaneous Breathing Test; Intensive Care Units (ICUs)
Keywords: Humidified high flow; Cardiac ultrasound; Spontaneous breathing trial; T-Piece

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The ultrasound evaluator will re-read and measure cardiac indexes on anonymized loops.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- EVS1-EVS2-EVS3 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial
- EVS1-EVS3-EVS2 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial
- EVS2-EVS3-EVS1 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial
- EVS2-EVS1-EVS3 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial
- EVS3-EVS1-EVS2 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial
- EVS3-EVS2-EVS1 (specific order of procedures) (Experimental): EVS1: Humidified High Flow Spontaneous Breathing Trial EVS2: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial EVS3: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial
  Interventions: Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial; Diagnostic Test: Pressure Support Spontaneous Breathing trial; Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial

INTERVENTIONS:
Diagnostic Test: No Pressure Support No Positive End Expiratory Pressure Spontaneous Breathing Trial — The spontaneous breathing test is carried out with the patient connected to the ventilator, reducing both the positive end-expiratory pressure (PEEP) and the pressure support to 0 cmH2O, for 15 minutes.
Diagnostic Test: Pressure Support Spontaneous Breathing trial — The spontaneous breathing test is carried out with the patient connected to the ventilator, reducing the positive end-expiratory pressure (PEEP) to 0 cmH2O and the pressure support to 7 cmH2O, for 15 minutes. A 10-minute washout period is left before the start of the next SBT modality.
Diagnostic Test: Humidified High Flow Spontaneous Breathing Trial — The spontaneous breathing trial is carried out with humidified high flow ventilator mode set at 50 liters per minute for 15 minutes. The patient will be connected to the ventilator via a specific connector enabling the administration of humidified high flow. A 10-minute washout period is left before the start of the next SBT modality.

SUMMARY:
The goal of this clinical trial is to evaluate the evolution of a cardiac ultrasound index (E/E') during 3 spontaneous breathing trials in Intensive Care Unit (ICU) adults (over 18 years) patients at risk for weaning failure. The main objective is to find out which spontaneous breathing trial is the least demanding in terms of heart work.

Investigators will compare 3 consecutive spontaneous breathing trials in a random order to see if one is superior to the others.

Participants will not have to perform any specific procedure apart from breathing without respiratory support during the spontaneous breathing trial. During these trials, the investigator will perform cardiac ultrasound measurements.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patient undergoing invasive mechanical ventilation for at least 24 hours and scheduled for a spontaneous breathing trial
* Richmond Agitation Sedation Scale (RASS) between -1 and +1
* Patient at high risk of re-intubation with at least one of the following criteria:

  * Underlying cardiac disease (left ventricular dysfunction with left ventricular ejection fraction ≤ 45%, documented ischemic heart disease, chronic atrial fibrillation, known history of cardiogenic pulmonary edema)
  * Underlying respiratory disease (COPD, Emphysema, bronchial dilatation, asthma, obesity/hypoventilation syndrome, restrictive lung disease)

Exclusion Criteria:

* Neuromuscular pathology (myasthenia type) preceding hospitalization
* Pregnant or breast-feeding women
* Patient already included in the study
* Protected person (under guardianship or curatorship)
* Person under court protection
* Person not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic evaluation of cardio E/E' index during 3 randomly assigned cross-over spontaneous breathing trials. | At the 5th minute from beginning of each spontaneous breathing trial (each breathing trial is 15 minutes)
  An evaluator at the patient's bed will use the cardiac ultrasound probe. The patient will be installed in a semi-seated position and the E/E' index will be measured over 3 successive cardiac cycles if the patient is in sinus rhythm, or 5 successive cycles if the patient is in atrial fibrillation. The measurement is taken at the 5th minute of each spontaneous breathing trial. The cross-over order of trials will be randomized.
  Once the cardiac ultrasound loops have been recorded, a blinded evaluator will read back the ultrasound images, and his or her measurement will be used for the primary evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Orleans, Orléans, France